CLINICAL TRIAL: NCT01634841
Title: Effect of Daily Ingestion of Walnuts for 2 Years on Age-related Cognitive Decline and Macular Degeneration in Healthy Elderly Subjects: A Randomized, Single Blind, Dual Center, Controlled Trial
Brief Title: Walnuts and Healthy Aging
Acronym: WAHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: University of Barcelona (Other); California Walnut Commission (Other)
Responsible Party: Principal Investigator, Joan Sabate,DrPH, MD, Principal Investigator, Chair, Department of Nutrition, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5120066; 670715-3833 (Other: Loma Linda University)
Record Dates: First submitted 2012-06-20; First posted 2012-07-06 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Age Related Cognitive Decline; Age Related Macular Degeneration
Keywords: walnuts; age related cognitive decline; age related macular degeneration; healthy elderly subjects
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Walnut group (Active Comparator): This group will have their habitual diet supplemented with 30 to 45g (1 to 1.5 oz) of walnuts daily.
  Interventions: Dietary Supplement: Walnuts
- Control group (Active Comparator): This group will eat their habitual diet and refrain from eating walnuts.
  Interventions: Other: habitual diet

INTERVENTIONS:
Dietary Supplement: Walnuts — 30 to 60g (1 to 2 oz) per day of walnuts
  Arms: Walnut group
Other: habitual diet — Dietary information will be provided
  Arms: Control group

SUMMARY:
This will be a systematic investigation of the role of walnuts in preventing or slowing age related cognitive decline and age related macular degeneration. 700 subjects will be recruited between 2 sites, Loma Linda University in California, USA and Hospital Clinic in Barcelona, Spain. Participants will be randomly assigned to either the walnut group or the control group for a 2 year intervention. Baseline and annual data will be collected and analyzed.

DETAILED DESCRIPTION:
Epidemiological studies suggest that nutrients such as n-3 polyunsaturated fatty acid, antioxidants and B-vitamins may protect against age related cognitive decline. Small human studies have shown beneficial effects of polyphenol rich foods on cognition and age related macular degeneration. Walnuts are a rich source of n-3 polyunsaturated fatty acid, alpha-linolenic acid, antioxidants, polyphenols and other bioactive compounds. A 2-year intervention will be conducted with healthy, elderly subjects to investigate the role of walnuts in preventing or slowing age related cognitive decline and age related macular degeneration.

350 subjects, age 63 to 79 years, will be recruited at each of 2 sites, Loma Linda University in California and Hospital Clinic in Barcelona. Participants will be randomly assigned to one of two groups: walnut group (habitual diet with 1 or 2 oz/d walnut supplement) or control group (habitual diet only). At baseline and yearly, cardiometabolic risk factors, red blood cell membrane fatty acids, urinary polyphenols and biomarkers of inflammation and oxidation will be measured. Eye exam, blood pressure and cognitive function tests will be measured at the beginning and end of 2 years. At the Barcelona site only, participants will be given a brain MRI and carotid ultrasound.

Descriptive results will be reported as mean plus/minus standard deviation. Primary analysis will be carried out on the basis of groups as randomly assigned. Results will be presented as appropriate effect sizes with a measure of precision (95% CI). Analysis of covariates gender, age, educational status will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* 63 to 79 years old
* healthy men and women
* able to attend clinic at a study sites

Exclusion Criteria:

* illiteracy or inability to understand the protocol
* unable to undergo neurophysiological tests
* morbid obesity (BMI greater than or equal to ≥ 40 kg/m2)
* uncontrolled diabetes (HbA1c>85)
* uncontrolled hypertension
* prior cerebrovascular accident
* any relevant psychiatric illness, including major depression
* advanced cognitive deterioration, dementia
* other neurodegenerative diseases (i.e. Parkinson's disease)
* any chronic illness expected to shorten survival (heart, liver, cancer, etc)
* bereavement in the first year of loss
* bad dentures unless fixable dental prostheses are used
* allergy to walnuts
* customary us of fish oil or flaxseed oil supplements
* eye related exclusion criteria

Ages: 63 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 708 (Actual)
Dates: Start 2012-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in global cognitive composite score | 2 years
  The composite score will be calculated using the scores from the tests listed below. We will calculate the standardized scores of each test as the score of each participant minus the group mean and divide by its standard deviation. The composite score is the mean of the standardized scores.
  The 12 tests are: Rey Auditory Verbal Learning Test (RAVLT), Rey-Osterrieth Complex Figure (ROCF), Semantic Fluency (Animals), Boston Naming Test (BNT), Visual Object and Space Perception Battery (VOSP), Block Design section from the Wechsler Adult Intelligence Scale (WAIS-III), Trail Making Test (TMT), FAS Word Fluency, Stroop Color Word Test, Symbol Digit Modalities Test (SMDT) Digit Span from the WAIS-III and Conners Continuous Performance Test (CPT-II).
Changes from baseline in macular degeneration | 2 years
  This will be assessed: by stereoscopic digitized color fundus images graded by International Classification System for Age-Related Maculopathy (score range. 0 to 4; the higher the score, the worse the condition); by optical coherence tomography (OCT) measurements of macular thickness (in µm); by optical coherence tomography (OCT) measurements of retinal nervous fiber layer thickness (in µm).

SECONDARY OUTCOMES:
Change from baseline in brain cortical thickness | 2 years
  Changes will be assessed by brain magnetic resonance imaging (MRI) on a randomly selected subset of participants. Only in Barcelona center. Unit of measure is mm2.
Change from baseline in voxel-based morphometry | 2 years
  Changes will be assessed by brain magnetic resonance imaging (MRI) using GM density maps on a randomly selected subset of participants. Only in Barcelona center. Unit of measure is GM density.
Change from baseline in white matter hyperintensity volumes | 2 years
  Changes will be assessed by brain magnetic resonance imaging (MRI) on a randomly selected subset of participants. Only in Barcelona center. Unit of measure is mL.
Change from baseline in perfusion arterial spin labeling | 2 years
  Changes will be assessed by brain magnetic resonance imaging (MRI) on a randomly selected subset of participants. Only in Barcelona center. Unit of measure is ml/100 g/min.
Changes from baseline in brain activation | 2 years
  Changes will be assessed by Functional MRI (fMRI) on a randomly selected subset of participants. Only in Barcelona center. There are no units of measure.

OTHER OUTCOMES:
Change in carotid Intima-media thickness (mm) | 2 years
  Changes will be assessed by high-resolution ultrasound. Only in Barcelona center.
Incidence of plaque presence in carotid artery (yes/no) | 2 years
  Changes will be assessed by high-resolution ultrasound. Only in Barcelona center.
Change in carotid atheroma plaque height (mm) | 2 years
  Changes will be assessed by high-resolution ultrasound. Only in Barcelona center.
Change in body mass index (kg/m2) | 2 years
  BMI will be calculated as weight in kilograms divided by height in metres squared
Change in waist circumference (cm) | 2 years
  Waist circumference will be measured to the nearest 0.5 cm by using an anthropometric tape midway between the lowest rib and at the iliac crest at minimal respiration
Change in total fat (g) | 2 years
  Changes will be assessed by Dual-energy X-ray absorptiometry. Only in Barcelona center.
Change in Total lean tissue (g) | 2 years
  Changes will be assessed by Dual-energy X-ray absorptiometry. Only in Barcelona center.
Change in fasting serum total cholesterol (mg/dL) | 2 years
  Fasting serum total cholesterol will be measured by a standard enzymatic method
Change in fasting serum LDL-cholesterol (mg/dL) | 2 years
  Fasting serum LDL-cholesterol will be estimated by the Friedewald formula
Change in fasting serum HDL-cholesterol (mg/dL) | 2 years
  Fasting serum HDL-cholesterol will be measured by a precipitation technique
Change in fasting serum triglycerides (mg/dL) | 2 years
  Fasting triglycerides will be measured by a standard enzymatic method
Change in serum brain-derived neurotrophic factor (pg/mL) | 2 years
  Assessed by ELISA
Change in serum soluble-Selectin (ng/mL) | 2 years
  Assessed by ELISA
Change in serum soluble-intercellular Adhesion Molecule 1 (ng/mL) | 2 years
  Assessed by ELISA
Change in serum soluble-vascular cell adhesion molecule 1 (ng/mL) | 2 years
  Assessed by ELISA
Change in serum amyloid A (ng/mL) | 2 years
  Assessed by ELISA
Change in serum granulocyte-macrophage colony-stimulating factor (pg/mL) | 2 years
  Assessed by ELISA
Change in serum interferon-gamma (pg/mL) | 2 years
  Assessed by ELISA
Change in serum interleukin-1beta (pg/mL) | 2 years
  Assessed by ELISA
Change in serum interleukin-6 (pg/mL) | 2 years
  Assessed by ELISA
Change in serum tumor necrosis factor alpha (pg/mL) | 2 years
  Assessed by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Joan Sabate, MD, DrPH, Principal Investigator — Chair, Department of Nutrition; Emilio Ros, MD, PhD, Principal Investigator — Director Lipid Clinic, Endocrinology & Nutrition Service
Locations (2):
- Loma Linda University, Department of Nutrition, Loma Linda, California, United States
- Hospital Clinic, University of Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Cofan M, Checa A, Serra-Mir M, Roth I, Valls-Pedret C, Lopez-Illamola A, Domenech M, Rajaram S, Lazaro I, Sabate J, Ros E, Wheelock CE, Sala-Vila A. A Walnut-Enriched Diet for 2 Years Changes the Serum Oxylipin Profile in Healthy Older Persons. J Nutr. 2024 Feb;154(2):395-402. doi: 10.1016/j.tjnut.2023.12.007. Epub 2023 Dec 9. PMID 38081585
- [Derived] Fjell AM, Sorensen O, Wang Y, Amlien IK, Baare WFC, Bartres-Faz D, Boraxbekk CJ, Brandmaier AM, Demuth I, Drevon CA, Ebmeier KP, Ghisletta P, Kievit R, Kuhn S, Madsen KS, Nyberg L, Sole-Padulles C, Vidal-Pineiro D, Wagner G, Watne LO, Walhovd KB. Is Short Sleep Bad for the Brain? Brain Structure and Cognitive Function in Short Sleepers. J Neurosci. 2023 Jul 12;43(28):5241-5250. doi: 10.1523/JNEUROSCI.2330-22.2023. Epub 2023 Jun 26. PMID 37365003
- [Derived] Nyberg L, Magnussen F, Lundquist A, Baare W, Bartres-Faz D, Bertram L, Boraxbekk CJ, Brandmaier AM, Drevon CA, Ebmeier K, Ghisletta P, Henson RN, Junque C, Kievit R, Kleemeyer M, Knights E, Kuhn S, Lindenberger U, Penninx BWJH, Pudas S, Sorensen O, Vaque-Alcazar L, Walhovd KB, Fjell AM. Educational attainment does not influence brain aging. Proc Natl Acad Sci U S A. 2021 May 4;118(18):e2101644118. doi: 10.1073/pnas.2101644118. PMID 33903255
- [Derived] Fjell AM, Sorensen O, Amlien IK, Bartres-Faz D, Brandmaier AM, Buchmann N, Demuth I, Drevon CA, Duzel S, Ebmeier KP, Ghisletta P, Idland AV, Kietzmann TC, Kievit RA, Kuhn S, Lindenberger U, Magnussen F, Macia D, Mowinckel AM, Nyberg L, Sexton CE, Sole-Padulles C, Pudas S, Roe JM, Sederevicius D, Suri S, Vidal-Pineiro D, Wagner G, Watne LO, Westerhausen R, Zsoldos E, Walhovd KB. Poor Self-Reported Sleep is Related to Regional Cortical Thinning in Aging but not Memory Decline-Results From the Lifebrain Consortium. Cereb Cortex. 2021 Mar 5;31(4):1953-1969. doi: 10.1093/cercor/bhaa332. PMID 33236064
- [Derived] Sorensen O, Brandmaier AM, Macia D, Ebmeier K, Ghisletta P, Kievit RA, Mowinckel AM, Walhovd KB, Westerhausen R, Fjell A. Meta-analysis of generalized additive models in neuroimaging studies. Neuroimage. 2021 Jan 1;224:117416. doi: 10.1016/j.neuroimage.2020.117416. Epub 2020 Oct 2. PMID 33017652
- [Derived] Hooper L, Martin N, Jimoh OF, Kirk C, Foster E, Abdelhamid AS. Reduction in saturated fat intake for cardiovascular disease. Cochrane Database Syst Rev. 2020 Aug 21;8(8):CD011737. doi: 10.1002/14651858.CD011737.pub3. PMID 32827219
- [Derived] Hooper L, Martin N, Jimoh OF, Kirk C, Foster E, Abdelhamid AS. Reduction in saturated fat intake for cardiovascular disease. Cochrane Database Syst Rev. 2020 May 19;5(5):CD011737. doi: 10.1002/14651858.CD011737.pub2. PMID 32428300
- [Derived] Sala-Vila A, Valls-Pedret C, Rajaram S, Coll-Padros N, Cofan M, Serra-Mir M, Perez-Heras AM, Roth I, Freitas-Simoes TM, Domenech M, Calvo C, Lopez-Illamola A, Bitok E, Buxton NK, Huey L, Arechiga A, Oda K, Lee GJ, Corella D, Vaque-Alcazar L, Sala-Llonch R, Bartres-Faz D, Sabate J, Ros E. Effect of a 2-year diet intervention with walnuts on cognitive decline. The Walnuts And Healthy Aging (WAHA) study: a randomized controlled trial. Am J Clin Nutr. 2020 Mar 1;111(3):590-600. doi: 10.1093/ajcn/nqz328. PMID 31912155
- [Derived] Bartres-Faz D, Gonzalez-Escamilla G, Vaque-Alcazar L, Abellaneda-Perez K, Valls-Pedret C, Ros E, Grothe MJ. Characterizing the Molecular Architecture of Cortical Regions Associated with High Educational Attainment in Older Individuals. J Neurosci. 2019 Jun 5;39(23):4566-4575. doi: 10.1523/JNEUROSCI.2370-18.2019. Epub 2019 Apr 8. PMID 30962275
- [Derived] Domenech M, Serra-Mir M, Roth I, Freitas-Simoes T, Valls-Pedret C, Cofan M, Lopez A, Sala-Vila A, Calvo C, Rajaram S, Sabate J, Ros E. Effect of a Walnut Diet on Office and 24-Hour Ambulatory Blood Pressure in Elderly Individuals. Hypertension. 2019 May;73(5):1049-1057. doi: 10.1161/HYPERTENSIONAHA.118.12766. PMID 30879358
- [Derived] Freitas-Simoes TM, Cofan M, Blasco MA, Soberon N, Foronda M, Corella D, Asensio EM, Serra-Mir M, Roth I, Calvo C, Valls-Pedret C, Casaroli-Marano RP, Domenech M, Rajaram S, Sabate J, Ros E, Sala-Vila A. The red blood cell proportion of arachidonic acid relates to shorter leukocyte telomeres in Mediterranean elders: A secondary analysis of a randomized controlled trial. Clin Nutr. 2019 Apr;38(2):958-961. doi: 10.1016/j.clnu.2018.02.011. Epub 2018 Feb 17. PMID 29478886
- [Derived] Rajaram S, Valls-Pedret C, Cofan M, Sabate J, Serra-Mir M, Perez-Heras AM, Arechiga A, Casaroli-Marano RP, Alforja S, Sala-Vila A, Domenech M, Roth I, Freitas-Simoes TM, Calvo C, Lopez-Illamola A, Haddad E, Bitok E, Kazzi N, Huey L, Fan J, Ros E. The Walnuts and Healthy Aging Study (WAHA): Protocol for a Nutritional Intervention Trial with Walnuts on Brain Aging. Front Aging Neurosci. 2017 Jan 10;8:333. doi: 10.3389/fnagi.2016.00333. eCollection 2016. PMID 28119602
- [Derived] Fernandez-Cabello S, Valls-Pedret C, Schurz M, Vidal-Pineiro D, Sala-Llonch R, Bargallo N, Ros E, Bartres-Faz D. White matter hyperintensities and cognitive reserve during a working memory task: a functional magnetic resonance imaging study in cognitively normal older adults. Neurobiol Aging. 2016 Dec;48:23-33. doi: 10.1016/j.neurobiolaging.2016.08.008. Epub 2016 Aug 20. PMID 27636672
- [Derived] Vaque-Alcazar L, Sala-Llonch R, Valls-Pedret C, Vidal-Pineiro D, Fernandez-Cabello S, Bargallo N, Ros E, Bartres-Faz D. Differential age-related gray and white matter impact mediates educational influence on elders' cognition. Brain Imaging Behav. 2017 Apr;11(2):318-332. doi: 10.1007/s11682-016-9584-8. PMID 27535872